CLINICAL TRIAL: NCT05240807
Title: Comprehensive Characterization of Coronary Atherosclerotic Disease Using Photon Counting- Detector Dual-source CT and Its Impact on Patient Management
Brief Title: Clinical Impact of Cardiac Photon Counting CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Cynthia McCollough, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-004933; R01EB028590-02 (NIH)
Record Dates: First submitted 2022-01-14; First posted 2022-02-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary CT Angiography; Cardiac Stress Imaging; Photon Counting CT; Cardiac CT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clinical Coronary CTA Cohort (Experimental): Subjects scheduled for a clinically indicated coronary CTA will receive a research contrast-enhanced coronary CT angiogram using photon-counting CT
  Interventions: Diagnostic Test: Photon counting computed tomography (PC-CT)
- Clinical Nuclear Medicine or MRI Cardiac Stress Test Cohort (Experimental): Subjects scheduled for a clinically indicated nuclear medicine or MRI cardiac stress test will receive a research contrast-enhanced coronary CT angiogram using photon-counting CT at rest and after administration of a cardiac stress agent
  Interventions: Diagnostic Test: Photon counting computed tomography (PC-CT)

INTERVENTIONS:
Diagnostic Test: Photon counting computed tomography (PC-CT) — Cardiac CT imaging will be performed using a newly developed CT scanner that uses photon-counting detectors and the results compared to those from conventional CT, MRI, or nuclear medicine imaging systems

SUMMARY:
The purpose of this research trial is to determine whether images taken using a Photon Counting Detector CT scanner (PCD-CT) after the patient has received a drug that makes the heart work harder provide clinically important information about the severity of suspected coronary artery disease compared to CT imaging performed without using the drug that causes the heart to work harder.

DETAILED DESCRIPTION:
This study will focus on demonstrating the benefits of PCD-CT for clinical indications and findings where the improved spatial and temporal resolution, decreased quantum and electronic noise, improved spectral imaging capabilities, and increased iodine signal are expected to benefit the diagnosis and characterization of CAD and myocardial perfusion defects.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for coronary artery cardiac CT imaging or nuclear medicine or MRI cardiac perfusion within the Department of Radiology or Cardiology.
* Patients who are able and willing to sign the informed consent will be enrolled
* Negative pregnancy test if subject is of child-bearing age (females of child-bearing potential will be screened for pregnancy using a urine pregnancy test, which will be administered by the unit study coordinator at no cost to the patient).

Exclusion Criteria:

* Patients unable to provide written informed consent
* Pregnancy
* eGFR ≤ 30
* History of prior moderate or severe contrast reaction includes: unresponsiveness, severe respiratory distress, convulsions, arrhythmia, cardiopulmonary distress, progressive angioedema, laryngeal edema, dyspnea, bronchospasm, symptomatic tachycardia, symptomatic bradycardia, hypotension, hypertensive crisis.
* Any history of required premedication prior to iodinated contrast administration.
* Patients that consent to participation but do not undergo their clinically-indicated, contrast-enhanced CT, or nuclear medicine or MR perfusion scanning for any reason (e.g., bad IV, infiltration, reaction, change in indication).
* Patients experiencing atrial fibrillation, premature ventricular contractions or other heart rhythm abnormalities
* Hospitalized patients or patients under care in the Emergency Department

Specific exclusion criteria only for participation in the cardiac stress test arm of this study (requiring administration of Regadenoson):

* Anything by mouth within three hours of the examination
* Known hypersensitivity to Regadenoson, Adenosine, or Dipyridamole.
* Active ongoing wheezing or poorly controlled asthma or COPD (hospitalized within last month or receiving treatment for flair within last month).
* Second (type I or II) or third degree atrioventricular (AV) block or sinus node dysfunction unless patient has functioning artificial pacemaker.
* Ingested greater than 4 oz. of caffeine within the last 12 hours.
* Currently experiencing unstable coronary syndrome.
* Uncontrollable seizures within the last 3 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in disease status or post-exam recommendations | Through completion of CT exam, approximately 1 day
  A sub-specialty trained cardiac radiologist and a sub-specialty trained cardiologist will compare qualitative and quantitative results from the photon counting CT scans to the clinically ordered CT, MRI, or nuclear medicine scan. Clinically important differences in findings and recommendations will be recorded to assess the overall clinical impact of using photon-counting CT to assess patients with potential coronary artery disease, especially patients with heavily calcified, stented, or high-risk plaques, or having myocardial perfusion defects. Our premise is that the established benefits of PCD-CT, used with a dual-source geometry and advanced noise reduction and material decomposition algorithms, will yield clinically important differences in imaging findings that will impact patient management decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia McCollough, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Boleyn Andrist, Eyota, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No